CLINICAL TRIAL: NCT03499002
Title: Teaching Medical Students How to Suture: Standard Simulation vs in Situ
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: study was discontinued
Sponsor: Memorial University of Newfoundland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: MUNChrystal
Record Dates: First submitted 2018-03-26; First posted 2018-04-17 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2018-04

CONDITIONS: Sutured Laceration; Laceration
Keywords: Simulation; Medical Students; In Situ Simulation
MeSH Terms: conditions — Lacerations

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Research assistant will be present when student randomly chooses which environment they will learn how to suture in. The principal investigator will be unaware of this randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simulation Lab (Experimental)
  Interventions: Other: Simulated Learning Environment
- ER in situ Simulation (Experimental)
  Interventions: Other: Simulated Learning Environment

INTERVENTIONS:
Other: Simulated Learning Environment — Intervention is the environment in which the medical student will learn to practice how to suture. The end goal is to determine the impact each environment has on their ability to learn the skill.
  Other Names: Simulation lab; ER in situ simulation

SUMMARY:
The purpose of this project is to compare in situ simulation with standard lab simulation. To do this, 30 pre-clinical medical students will be randomized into the lab or ER and taught how to suture a simple laceration. To do this, a synthesized 'skin' will be placed over a volunteer's arm and will have an incision of a predetermined length.

DETAILED DESCRIPTION:
For this study, 30 first and second year students will be equally randomized to either a standard simulation lab or the ER department to learn the skill of suturing. These students will not have any knowledge of suturing prior to this study. Each group will have 15 students. Each student will be given access to the same suturing learning video. They will each attempt 15 sutures on a lab generated skin placed over a volunteer's arm. Each incision length will be predetermined and of the same length. The student will have the opportunity to re-watch the video in between each suture attempt. The volunteer will record the student's number of attempts and whether or not they had to review the video. The idea behind this, is that students should began to plateau with their learning after about 8-9 attempts and most will no longer require the video beyond that.After the 15 attempts, the student will immediately practice 6 sutures on a second skin over the volunteer's arm, again of a predetermined incision length. At this point the students will only be allowed to practice the suturing skill and will not have access to the learning video. At this point, the student's hands will be video recorded to assess the accuracy of the skill.One week after the learning session, regardless of the environment they initially learned in, the student will be brought to the ER and again allowed to practice 6 sutures on a simulated skin placed over a volunteer's arm. The incision will be the same length as the incision in the previous practice session. Again, the student's hands will be video recorded while practicing the 6 sutures.Afterward, the student will be given a questionnaire regarding which environment they practiced in and how prepared they felt to practice in the insitu environment without learning aids.

ELIGIBILITY:
Inclusion Criteria:

* Pre clinical medical students (year one or two)

Exclusion Criteria:

* Medical students not in first or second year training
* Extensive knowledge or background with suturing

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-04 (Estimated); Primary Completion 2018-05 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
How each simulated learning environment effects a student's ability to learn how to suture | 1 week
  Each student will complete a post survey questionnaire after their attempt to suture in the ER department. This will help determine the impact and therefore, which environment was more conducive to learning how to suture.

CONTACTS AND LOCATIONS:
Overall Officials: Chrystal Horwood, MD, Principal Investigator — Memorial University of Newfoundland and Labrador

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Roussin CJ, Weinstock P. SimZones: An Organizational Innovation for Simulation Programs and Centers. Acad Med. 2017 Aug;92(8):1114-1120. doi: 10.1097/ACM.0000000000001746. PMID 28562455
- [Result] Jagneaux T, Caffery TS, Musso MW, Long AC, Zatarain L, Stopa E, Freeman N, Quin CC, Jones GN. Simulation-Based Education Enhances Patient Safety Behaviors During Central Venous Catheter Placement. J Patient Saf. 2021 Sep 1;17(6):425-429. doi: 10.1097/PTS.0000000000000425. PMID 28984729
- [Result] Sorensen JL, Ostergaard D, LeBlanc V, Ottesen B, Konge L, Dieckmann P, Van der Vleuten C. Design of simulation-based medical education and advantages and disadvantages of in situ simulation versus off-site simulation. BMC Med Educ. 2017 Jan 21;17(1):20. doi: 10.1186/s12909-016-0838-3. PMID 28109296
- [Result] Ullman E, Kennedy M, Di Delupis FD, Pisanelli P, Burbui AG, Cussen M, Galli L, Pini R, Gensini GF. The Tuscan Mobile Simulation Program: a description of a program for the delivery of in situ simulation training. Intern Emerg Med. 2016 Sep;11(6):837-41. doi: 10.1007/s11739-016-1401-2. Epub 2016 Feb 9. PMID 26861702
- [Result] Haji FA, Rojas D, Childs R, de Ribaupierre S, Dubrowski A. Measuring cognitive load: performance, mental effort and simulation task complexity. Med Educ. 2015 Aug;49(8):815-27. doi: 10.1111/medu.12773. PMID 26152493
- [Result] Rosen MA, Hunt EA, Pronovost PJ, Federowicz MA, Weaver SJ. In situ simulation in continuing education for the health care professions: a systematic review. J Contin Educ Health Prof. 2012 Fall;32(4):243-54. doi: 10.1002/chp.21152. PMID 23280527
- [Result] Petrosoniak A, Auerbach M, Wong AH, Hicks CM. In situ simulation in emergency medicine: Moving beyond the simulation lab. Emerg Med Australas. 2017 Feb;29(1):83-88. doi: 10.1111/1742-6723.12705. Epub 2016 Oct 17. PMID 27748042
- [Result] Naismith LM, Cheung JJ, Ringsted C, Cavalcanti RB. Limitations of subjective cognitive load measures in simulation-based procedural training. Med Educ. 2015 Aug;49(8):805-14. doi: 10.1111/medu.12732. PMID 26152492